CLINICAL TRIAL: NCT02145780
Title: Polyphenols: Protection From Overfeeding-induced Insulin Resistance?
Brief Title: Polyphenols and Overfeeding
Acronym: Poly-Nut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2013-807
Record Dates: First submitted 2014-05-13; First posted 2014-05-23 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Overfeeding
Keywords: Overfeeding; Fat distribution; Subcutaneous and visceral adipose tissue; Insulin sensitivity; Insulin resistance; Peripheral and hepatic insulin sensitivity; Stable isotopes; Lipid oxidation; Energy expenditure; Muscle and subcutaneous adipose tissue gene expression
MeSH Terms: conditions — Insulin Resistance | interventions — Dietary Supplements; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2g of grape polyphenol extract supplement (Experimental): Men will have to consume daily 2g of grape polyphenol extract during the 31 days of overfeeding.
  Interventions: Dietary Supplement: 2g of grape polyphenol extract
- 2g of placebo (lactose) (Placebo Comparator): Men will have to consume daily 2g of placebo during the 31 days of overfeeding.
  Interventions: Dietary Supplement: Dietary Supplement: 2g of placebo (lactose)

INTERVENTIONS:
Dietary Supplement: 2g of grape polyphenol extract — Men will have to consume daily 2g of grape polyphenol extract during the 31 days of overfeeding.
  Arms: 2g of grape polyphenol extract supplement
Dietary Supplement: Dietary Supplement: 2g of placebo (lactose) — Men will have to consume daily 2g of placebo during the 31 days of overfeeding.
  Arms: 2g of placebo (lactose)

SUMMARY:
Obesity is a complex and multifactorial disease representing a major public health challenge. Indeed, overweight and obese people carry a major risk of developing insulin resistance and type 2 diabetes mellitus. It has been demonstrated that polyphenols could be used to counteract some of the mechanisms involved in the generation of insulin resistance. The model of overfeeding represents a very good study model of the metabolic complications of obesity, since it has been shown to induce a transient state of insulin resistance in the human.

The purpose of this research is to study the effects of a overfeeding (+50% of daily caloric needs over 31 days) with or without polyphenols supplementation (2g/days over 31 days) on insulin sensitivity measured in the setting of a hyperinsulinemic euglycemic clamp and on post prandial partitioning of exogenous lipids after a test meal.

During 31 days, the volunteers will consume chocolate bars, chips, chocolate breads and cola in addition to their usual diet and will be supplemented with 2g of grape polyphenols extract or with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged from 18 to 55 years
* Body Mass Index of 23 to 27 kg/m²
* Normal blood pressure
* Fasting glycemia < 7 mmol/L
* CRPus < 10mg/L
* Triglycerides ≤ 3mmol/L

Exclusion Criteria:

* Medical or surgical history which may affect the results (renal -cardiovascular - hepatic- endocrine-inflammatory diseases)
* Subjects under treatment which may interfere with the measured parameters
* Eating disorder
* Intensive sportive activity
* Dairy products allergy or intolerance

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Peripheral insulin sensitivity | During 31 days
  Volunteers will have peripheral and hepatic insulin sensitivity determined by using a two-stage hyperinsulinemic euglycemic clamp with stable isotopically labeled tracer infusion.

SECONDARY OUTCOMES:
Hepatic insulin sensitivity | before and after the 31 days of overfeeding
  Endogenous glucose production (EGP) will be determined during the last 30 minutes of the low-dose insulin infusion.
Change in genes expression in adipose and muscle tissues | Before and after the 31 days of overfeeding
  RT-PCR
Anthropometry, Fat quantification and Abdominal fat distribution | During 31 days
  Weight, height, waist and hip circumferences, fat mass using dual x-ray absorptiometry (DEXA) and abdominal fat distribution using resonance magnetic imaging (RMI).
Fasting and Postprandial partitioning of exogenous lipid | Fasting and during all the postprandial period (0-300 minutes)
  13C enrichment will be measured in blood samples and breath test during a test meal performed before and after the 31 days of overfeeding.
Modification in intestinal microbiota | Before and after the 31 days of overfeeding
  Feces analyses
Energy expenditure and substrate oxidation with indirect calorimetry | Fasting and during all the postprandial period (0-300 minutes)
  Energy metabolism will be measured before and after the 31 days of overfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, MD, PhD, Principal Investigator — Rhône Alpes Human Nutrition Center (CRNH Rhône-Alpes)
Locations (1):
- Rhône Alpes Human Nutrition Center (CRNH Rhône-Alpes), Pierre-Bénite, France

REFERENCES:
- [Derived] Bartova S, Madrid-Gambin F, Fernandez L, Carayol J, Meugnier E, Segrestin B, Delage P, Vionnet N, Boizot A, Laville M, Vidal H, Marco S, Hager J, Moco S. Grape polyphenols decrease circulating branched chain amino acids in overfed adults. Front Nutr. 2022 Oct 26;9:998044. doi: 10.3389/fnut.2022.998044. eCollection 2022. PMID 36386937
- [Derived] Segrestin B, Delage P, Nemeth A, Seyssel K, Disse E, Nazare JA, Lambert-Porcheron S, Meiller L, Sauvinet V, Chanon S, Simon C, Ratiney H, Beuf O, Pralong F, Yassin NA, Boizot A, Gachet M, Burton-Pimentel KJ, Vidal H, Meugnier E, Vionnet N, Laville M. Polyphenol Supplementation Did Not Affect Insulin Sensitivity and Fat Deposition During One-Month Overfeeding in Randomized Placebo-Controlled Trials in Men and in Women. Front Nutr. 2022 May 9;9:854255. doi: 10.3389/fnut.2022.854255. eCollection 2022. PMID 35614978